CLINICAL TRIAL: NCT03037242
Title: Multi-Center Prospective Clinical and Radiographic Outcomes of Meniscus Root Repair Using a Transtibial Pullout Technique
Brief Title: Outcomes of Meniscus Root Repair Using a Transtibial Pullout Technique
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel B. F. Saris, Professor of Orthopedics, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-005841
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transtibial pullout technique (Other): Evaluation of the clinical and radiographic outcomes for patients undergoing a meniscus root repair (MRR) using a transtibial pullout technique.
  Interventions: Procedure: Transtibial pullout technique

INTERVENTIONS:
Procedure: Transtibial pullout technique — Evaluating radographs

SUMMARY:
The results of this study will optimize the care for patients with a meniscus root tear. Surgeons will be able to determine if MRR (meniscus root repair) with transtibial pullout technique is an effective treatment and will identify potential risk factors for poor clinical outcomes. In addition, investigators will determine if MRR is successful in delaying the radiographic progression of arthritis in the involved compartment.

DETAILED DESCRIPTION:
The loss of attachment at the root of the meniscus impairs the ability to maintain hoop strain when the tibiofemoral joint is loaded. This loss of hoop strain is responsible for the increased pressure on the articular cartilage.

This new awareness has prompted surgeons to consider surgical repair for treatment of meniscal root avulsions. Despite this recent focus on results of surgical repair, prospective studies are lacking, and the optimal surgical indications and technique have not been optimized.

ELIGIBILITY:
Inclusion Criteria:

1. Meniscus root avulsion tear (defined as meniscus posterior horn root avulsion or full thickness tear within 9 mm of the root attachment)
2. Age 18-65
3. Ligament injury with concomitant reconstruction is acceptable
4. Malalignment with corrective osteotomy is acceptable

Exclusion Criteria:

1. Subchondral collapse on pre-op MRI
2. Extrusion greater than 3 mm
3. Intra-op Outerbridge grade 3 or greater chondromalacia
4. Intra-op poor quality meniscus tissue
5. Mal-alignment greater than 5 degrees without corrective osteotomy
6. Obesity with BMI over 40
7. Kellgren Lawrence > grade 2
8. Worker's compensation status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Tegner activity score | baseline, 2 years
  Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury. The score varies from 0-10.
  A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports >6 score can only be achieved if the person participates in recreational or competitive sport.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Saris, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Columbia Orthopaedic Group, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krych AJ, Song BM, Nauert RF 3rd, Cook CS, Levy BA, Camp CL, Stuart MJ, Smith PA. Prospective Consecutive Clinical Outcomes After Transtibial Root Repair for Posterior Meniscal Root Tears: A Multicenter Study. Orthop J Sports Med. 2022 Feb 24;10(2):23259671221079794. doi: 10.1177/23259671221079794. eCollection 2022 Feb. PMID 35237699
- [Derived] Krych AJ, Nauert RF 3rd, Song BM, Cook CS, Johnson AC, Smith PA, Stuart MJ. Association Between Transtibial Meniscus Root Repair and Rate of Meniscal Healing and Extrusion on Postoperative Magnetic Resonance Imaging: A Prospective Multicenter Study. Orthop J Sports Med. 2021 Aug 16;9(8):23259671211023774. doi: 10.1177/23259671211023774. eCollection 2021 Aug. PMID 34423058
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials